CLINICAL TRIAL: NCT02761369
Title: Comparison of Two Deep TMS Protocols With Paired Associative Stimulation (PAS) for the Treatment of Food Addiction in Severe Obesity
Brief Title: Deep Transcranial Magnetic Stimulation (TMS) With Paired Associative Stimulation (PAS) for the Treatment of Food Addiction in Obesity
Acronym: FAOB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOR-0324-15-CTIL
Record Dates: First submitted 2016-04-20; First posted 2016-05-04 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: food addiction; obesity; deep TMS; PAS; Food Stroop; brain laterality; EEG; INP
MeSH Terms: conditions — Obesity; Food Addiction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A PAS protocol, right-to-left, via deep TMS (Experimental): Via a multi-channel deep TMS device with an H-coil (Brainsway Ltd), a PAS protocol, starting with the right DLPFC
  Interventions: Device: A multi-channel deep TMS device with an H-coil (Brainsway Ltd)
- A PAS protocol, left-to-right, via deep TMS (Experimental): Via a multi-channel deep TMS device with an H-coil (Brainsway Ltd), a PAS protocol, starting with the left DLPFC
  Interventions: Device: A multi-channel deep TMS device with an H-coil (Brainsway Ltd)
- A sham PAS protocol, via deep TMS (Sham Comparator): Via a multi-channel deep TMS device with an H-coil (Brainsway Ltd), a sham PAS protocol, starting with the right DLPFC (@ 40% of individual MT)
  Interventions: Device: A multi-channel deep TMS device with an H-coil (Brainsway Ltd)

INTERVENTIONS:
Device: A multi-channel deep TMS device with an H-coil (Brainsway Ltd) — A 3-week long treatment (15 days). Treatment session consist of 300 rapidly occurring pairs of pulses over the dorsolateral prefrontal cortex (at a frequency of 10 Hz and intensity of 110% of individual's motor threshold), with a 5-seconds interval, for a duration of 1800 seconds in total.

SUMMARY:
The neurobiological underpinnings of obesity point to brain asymmetry in cortical and deeper brain regions. Furthermore, chemical, structural and functional imbalance in cortical and sub-cortical brain regions alters reward processing, attentional control and self-regulation in food-addicted obese individuals. In this study the investigators use TMS with a special multichannel H-coil developed by their lab to safely stimulate cortical and deeper brain regions in obese humans. The investigators aim to produce interhemispheric neuroplasticity (INP) using a paired associative stimulation (PAS) protocol over the DLPFC, to restore neurobiological functioning, alleviate food addiction symptoms, and promote weight loss.

ELIGIBILITY:
Inclusion Criteria:

* 30 ≤ BMI ≥ 40.
* Having had at least one prior conventional weight loss attempt, but no current weight loss attempts or over the last 3 months.
* Having satisfied a safety screening questionnaire for TMS (Keel, 2001)
* Omnivorous
* Have not had experience with TMS of any kind

Exclusion Criteria:

* The participant experiences tremor in any limb.
* The participant experiences seizures.
* The participant has a history of epilepsy or seizure (EXCEPT those therapeutically induced by ECT), or a history of such in first degree relatives.
* The participant is at increased risk for seizures for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or a history of significant head trauma with loss of consciousness for > 5 minutes.
* The participant has a history of head injury.
* The participant suffers from an unstable physical disease, such as high blood pressure (>150 mmHg systolic / diastolic > 110 mmHg) or acute, unstable cardiac disease The participant is at a high risk for severe violence or suicidal tendencies, assessed during the screening interview (see appendix 4).
* The participant has metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neuro-stimulators, intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* The participant is having, or has had, any metal in the head (outside the mouth).
* The participant suffers from a significant neurological disorder or insult including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure
  * Space occupying brain lesion
  * History of cerebrovascular accident
  * Transient ischemic attack within the last two years
  * Cerebral aneurysm
  * Dementia
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
* The participant has any cognitive or functional disability, according to criteria specified in the DSM-V, such as active psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-V; Axis I and Axis II) diagnosed within the last year.
* The participant has started or changed a psychotropic prescription within the last three months.
* The participant has current alcohol or other substance abuse or dependence, or has had one over the last 12 months prior to recruitment.
* The participant can't reliably communicate with the investigator, or is unlikely to cope with the requirements of the experiment.
* The participant is having a known or suspected pregnancy or lactation.
* The participant is a sexually-active woman of childbearing age, who does not use a medically accepted form of contraception.
* The motor threshold can't be found or quantified.
* The PI decides that the participant should be withdrawn from the study for the safety and welfare of the participant. For example, the participant experiences adverse event which is contraindicated with the continuation in the study.
* A history of intolerance to a TMS treatment.
* The participant asks for withdrawal

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-18 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Change in weight between baseline versus the end of the treatment (day 15) and follow-up (a month after day 15)
  Unit of measure: BMI in kg/m^2 (weight in kilograms, height in meters)

SECONDARY OUTCOMES:
Performance on a food Stroop test | Change in performance between baseline versus the end of the treatment (day 15) and follow-up (a month after day 15)
  Unit of measure: reaction time (in milliseconds)
Food addiction symptoms | Change between baseline versus the end of the treatment (day 15) and follow-up (a month after day 15)
  Yale Food Addiction Scale (YFAS)
Safety and tolerability of a PAS protocol using the multi-channel deep TMS system, measured via the number of adverse events (AE) | Throughout the study period, estimated as 2 years
  Measured via the number of adverse events
Eating behavior (cognitive restraint, disinhibition, and hunger) | Change between baseline versus the end of the treatment (day 15) and follow-up (a month after day 15)
  Three Factor Eating Questionnaire (TFEQ)
Quality of life | Change between baseline and the end of the treatment (day 15) and follow-up (a month after day 15)
  Health Status Scale Short-form 36 (SF-36)
Implementation of INP | Changes in cortical excitability between baseline versus following 15 days of treatment
  1. Acute change in INP, assessed via changes in cortical excitability (measured via EEG and TCI) between pre- and post PAS administration. 2. Chronic change in INP assessed as change in cortical excitability between baseline versus the end of the treatment (day 15) and follow up (measured via EEG and TCI)

OTHER OUTCOMES:
General mood | Change between baseline versus the end of the treatment (day 15) and follow-up (a month after day 15)
  Positive Affect Negative Affect Schedule (PANAS)

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Avinoach, MD, Principal Investigator — Soroka UMC; Roni Aviram-Friedman, PhD, Study Director — Ben-Gurion University of the Negev; Abraham Zangen, PhD, Study Chair — Ben-Gurion University of the Negev
Locations (1):
- SorokaUMC, Beersheba, Israel